CLINICAL TRIAL: NCT05442086
Title: Music and Auditory Beat Stimulation and Its Effect on Anxiety
Brief Title: Music and ABS as a Potential Anxiety Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Frank Russo, Professor, Toronto Metropolitan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-068 LUCiD Anxiety
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music and Theta Auditory Beat Stimulation (Experimental): Behavioural: Listening to calm music and auditory beat stimulation Participants will listen to calm music with theta auditory beat stimulation for 24-27 minutes
  Interventions: Behavioral: Music and Theta Auditory Beat Stimulation
- Pink Noise (control) (Sham Comparator): Behavioural: Listening to pink noise Participants will listen to pink noise for 24 minutes
  Interventions: Behavioral: Pink Noise (control)

INTERVENTIONS:
Behavioral: Music and Theta Auditory Beat Stimulation — Participants will listen to calm music with theta auditory beat stimulation for 24-27 minutes
  Arms: Music and Theta Auditory Beat Stimulation
Behavioral: Pink Noise (control) — Participants will listen to pink noise for 24 minutes
  Arms: Pink Noise (control)

SUMMARY:
Anxiety is a growing problem and has been steadily increasing, particularly in the adolescent and young adult populations in the past 24 years. Music and auditory beat stimulation (ABS) in the theta frequency range (4-7 Hz) are sound-based anxiety treatments that have been investigated in prior studies with subjective measures of anxiety. Here, the anxiety-reducing potential of calm music combined with theta ABS will be examined in a large sample of participants with objective psychophysiological measures (heart rate variability and EEG), stress hormone measures (salivary cortisol) along with subjective measures (STICSA state). Participants with a GAD-2 score of 1 or higher (indicating generalized anxiety) will be randomly assigned to a single 24-27 minute session of sound-based treatment: combined (music & ABS), or pink noise (control). Pre- and post-intervention heart rate variability and EEG band power (alpha, beta, delta, and theta bands), salivary cortisol, along with somatic and cognitive state anxiety measures (STICSA State) will be collected along with trait anxiety (STICSA Trait), and music absorption (Absorption in Music Scale). The investigators predict that the music & ABS condition will have significantly increased power in the theta and alpha bands, higher heart rate variability, higher state anxiety reduction, and lower salivary cortisol levels compared to the pink noise control condition.

DETAILED DESCRIPTION:
In this study, the investigators will examine and compare the effectiveness of a combination of music and theta auditory beat stimulation (ABS) (as measured by the State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA)) compared to a control condition (pink noise). Prior work has demonstrated that ABS and music both reduce anxiety when presented on their own. It is hypothesized that music with ABS will lead to significantly lower anxiety levels and increased calmness compared to the pink noise control condition. Approximately 50 participants with a GAD-2 score of 1 or more (indicating generalized anxiety) will be recruited from the greater Toronto area. The study will be conducted in the SMART lab at Toronto Metropolitan University and the experimental treatment will be presented through earphones connected to a laptop. Upon arrival in the lab research staff will go over experimental expectations, and participants will be asked to fill out the Absorption in Music Scale (AIMS), the Positive and Negative Affect Scale (PANAS), and Self-Assessment Manikin (SAM), and the STICSA trait and state. They will also be asked if they take any medication or use any alternative techniques to manage their anxiety (Anxiety Coping Measures Questionnaire). A baseline salivary cortisol sample will be taken from participants. Participants will then undergo EEG administration, assessment of spontaneous blink rate, and HRV, first obtaining a baseline level of these measures. EEG (alpha, beta, delta, and theta bands) will be recorded using the BioSemi EEG system via 64 scalp electrode sites according to the international 10-20 electrode system as done in a previous study examining EEG response to meditation. Linked mastoids will serve as a reference. Horizontal eye movements will be recorded using two electrodes placed 1 cm lateral to the outer canthi of each eye. Vertical eye movement potentials will be recorded using two electrodes placed in the center of the supraorbital and infraorbital regions of the left eye. These will be used to obtain the spontaneous blink rate of participants which is an analog of the sensitivity and responsiveness of the mesostriatal dopaminergic system that has in previous studies determined the degree to which gamma binaural beats affect cognition. Heart rate variability will also be recorded via the BioSemi system with two flat active electrodes attached to the participant's left and right wrists. Participants will then listen to their randomly assigned intervention for 24-27 minutes (music with theta ABS or pink noise). A post-intervention salivary cortisol sample will be taken along with a post-intervention EEG and HRV reading and the completion of the STICSA state anxiety questionnaire. An additional salivary cortisol sample will be taken 15 minutes after the end of the auditory treatment. The investigators predict that the music & ABS condition will have significantly increased power in the theta and alpha bands compared to the pink noise control condition. The investigators also predict that the music & ABS condition will have higher heart rate variability compared to the pink noise control condition. The investigators also expect to see significantly higher state anxiety reduction and significantly lower salivary cortisol levels in the music & ABS condition compared to the pink noise control condition.

ELIGIBILITY:
Inclusion Criteria:

* GAD-2 score of 1 or higher indicating generalized anxiety.
* Age between 18-30 years
* Undergraduate student
* Comfortable speaking and understanding English
* Self-reported normal hearing

Exclusion Criteria:

* Self-reported history of cardiovascular conditions (e.g., arrhythmia, heart disease)
* History of seizures or epilepsy

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Anxiety: EEG band power (alpha, beta, delta and theta bands) | 24-27 minutes
  EEG band power is a good objective physiological measure of anxiety and relaxation. It has good reliability and validity and has been used as an anxiety/relaxation measure in multiple studies (Aftanas, Pavlov, Reva, & Varlamov, 2003; Gálvez, Recuero, Canuet, & Del-Pozo, 2018; Knyazev, Savostyanov, & Levin, 2005; Lee, Bhattacharya, Sohn, & Verres, 2012; Tarrant, Viczko, & Cope, 2018).
Anxiety: Heart rate variability (HRV) | 24-27 minutes
  Heart rate variability is a good objective physiological measure of anxiety. It has good reliability and validity and has been used as an anxiety measure in multiple studies (Chalmers, Quintana, Abbott, & Kemp, 2014; Gorman & Sloan, 2000; Licht, de Geus, van Dyck, & Penninx, 2009; Pittig, Arch, Lam, & Craske, 2013).
Anxiety: Stress hormone levels: Salivary cortisol | 24-27 minutes
  Salivary cortisol is a good objective measure of stress and anxiety. It has good reliability and validity and has been used as an anxiety measure in multiple studies (Mantella et al., 2008; Vedhara et al., 2003; Vreeburg et al., 2010).
Anxiety: State Trait Inventory for Cognitive and Somatic Anxiety (STICSA) | 24-27 minutes
  The State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA) is a 21-item measure designed to measure somatic (11 items) and cognitive symptoms (10 items) of anxiety at both the trait and state levels. To differentiate between state and trait anxiety symptoms, participants will complete two versions of the measure, one where they rate how they "feel right now at this very moment" (STICSA-State) and one where they rate "how they feel in general" (STICSA-Trait). Respondents rate the degree to which each item is true for them on a Likert scale ranging from 1 = not at all to 4 = very much so. Scores on the STICSA can range from 10 - 40 (cognitive) or 11 - 44 (somatic), with higher scores indicating greater anxiety.
Self-Assessment Manikin | 24-27 minutes
  Two series of Self-Assessment Manikins (SAM) will be administered to assess state emotional valence and arousal before and after the audio intervention. Participants will be asked to rate on two scales with accompanying images how they are feeling right now (unhappy to happy) and their energy levels from calm to excited both on a scale from 1-5. The pre-intervention SAM serves two purposes: the first, to assess baseline affect and the second, to select the playlist that the participant listens to if assigned to the audio intervention. The post-intervention SAM will serve to assess changes in affect following the intervention.

SECONDARY OUTCOMES:
Mood: Positive and Negative Affect Scale (PANAS) | 24-27 minutes
  The PANAS has good reliability and validity and has been widely used in many studies to assess mood (Gray, 2007; Watson, Clark, & Tellegen, 1988). This scale generates two scores: 1) Positive affect (higher score indicates a better outcome), scores range from 10-50. 2) Negative affect (higher score indicates worse outcome), scores range from 10-50.
Absorption in Music Scale (AIMS) | 24-27 minutes
  The Absorption in Music Scale (AIMS) is a 34-item measure of individuals' ability and willingness to allow music to draw them into an emotional experience. The Absorption in Music Scale (AIMS) was administered post-intervention, after completing all other post-intervention measures to avoid biasing responses. The AIMS will serve as a sub-group analysis to assess if individuals who report higher absorption respond better to the audio intervention in the treatment condition. The AIMS demonstrates strong convergent validity with the Tellegen Absorption Scale (r = .76) and the Musical Involvement Scale (r = .74).
Anxiety Coping Measures | 24-27 minutes
  This is a self-made questionnaire which asks whether the participant takes any anxiety medications, and about other coping strategies they may already employ.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Russo, PhD, Principal Investigator — Toronto Metropolitan University (formerly Ryerson University)
Locations (1):
- Toronto Metropolitan University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data for EEG band power, Heart rate variability (HRV), salivary cortisol, STICSA state anxiety, and PANAS measures will be shared on the Open Science Framework.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available on the Open Science Framework (osf.io) when the pre-print of the study is uploaded to PsyArXiv. After that point the data will be available for a period of 5 years.
Access Criteria: All supporting information will be publicly accessible on the Open Science Framework (osf.io).

REFERENCES:
- [Background] Aftanas LI, Pavlov SV, Reva NV, Varlamov AA. Trait anxiety impact on the EEG theta band power changes during appraisal of threatening and pleasant visual stimuli. Int J Psychophysiol. 2003 Nov;50(3):205-12. doi: 10.1016/s0167-8760(03)00156-9. PMID 14585489
- [Background] Bados A, Gomez-Benito J, Balaguer G. The state-trait anxiety inventory, trait version: does it really measure anxiety? J Pers Assess. 2010 Nov;92(6):560-7. doi: 10.1080/00223891.2010.513295. PMID 20954057
- [Background] Bringman H, Giesecke K, Thorne A, Bringman S. Relaxing music as pre-medication before surgery: a randomised controlled trial. Acta Anaesthesiol Scand. 2009 Jul;53(6):759-64. doi: 10.1111/j.1399-6576.2009.01969.x. Epub 2009 Apr 14. PMID 19388893
- [Background] Chalmers JA, Quintana DS, Abbott MJ, Kemp AH. Anxiety Disorders are Associated with Reduced Heart Rate Variability: A Meta-Analysis. Front Psychiatry. 2014 Jul 11;5:80. doi: 10.3389/fpsyt.2014.00080. eCollection 2014. PMID 25071612
- [Background] Davis, W. B., & Thaut, M. H. (1989). The Influence of Preferred Relaxing Music on Measures of State Anxiety, Relaxation, and Physiological Responses. Journal of Music Therapy, 26(4), 168-187. doi:10.1093/jmt/26.4.168
- [Background] Galvez G, Recuero M, Canuet L, Del-Pozo F. Short-Term Effects of Binaural Beats on EEG Power, Functional Connectivity, Cognition, Gait and Anxiety in Parkinson's Disease. Int J Neural Syst. 2018 Jun;28(5):1750055. doi: 10.1142/S0129065717500551. Epub 2017 Nov 13. PMID 29297265
- [Background] Gorman JM, Sloan RP. Heart rate variability in depressive and anxiety disorders. Am Heart J. 2000 Oct;140(4 Suppl):77-83. doi: 10.1067/mhj.2000.109981. PMID 11011352
- [Background] Gray, E. K., Watson, D. (2007). Assessing positive and negative affect via self-report. In J. A. Coan, Allen, J.J.B. (Ed.), Handbook of emotion elicitation and assessment. New York, NY: Oxford University Press.
- [Background] Gros DF, Antony MM, Simms LJ, McCabe RE. Psychometric properties of the State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA): comparison to the State-Trait Anxiety Inventory (STAI). Psychol Assess. 2007 Dec;19(4):369-81. doi: 10.1037/1040-3590.19.4.369. PMID 18085930
- [Background] Isik BK, Esen A, Buyukerkmen B, Kilinc A, Menziletoglu D. Effectiveness of binaural beats in reducing preoperative dental anxiety. Br J Oral Maxillofac Surg. 2017 Jul;55(6):571-574. doi: 10.1016/j.bjoms.2017.02.014. Epub 2017 Mar 18. PMID 28325532
- [Background] Jongkees BJ, Colzato LS. Spontaneous eye blink rate as predictor of dopamine-related cognitive function-A review. Neurosci Biobehav Rev. 2016 Dec;71:58-82. doi: 10.1016/j.neubiorev.2016.08.020. Epub 2016 Aug 21. PMID 27555290
- [Background] Knyazev GG, Savostyanov AN, Levin EA. Uncertainty, anxiety, and brain oscillations. Neurosci Lett. 2005 Oct 28;387(3):121-5. doi: 10.1016/j.neulet.2005.06.016. PMID 16002215
- [Background] Lagopoulos J, Xu J, Rasmussen I, Vik A, Malhi GS, Eliassen CF, Arntsen IE, Saether JG, Hollup S, Holen A, Davanger S, Ellingsen O. Increased theta and alpha EEG activity during nondirective meditation. J Altern Complement Med. 2009 Nov;15(11):1187-92. doi: 10.1089/acm.2009.0113. PMID 19922249
- [Background] Lee EJ, Bhattacharya J, Sohn C, Verres R. Monochord sounds and progressive muscle relaxation reduce anxiety and improve relaxation during chemotherapy: a pilot EEG study. Complement Ther Med. 2012 Dec;20(6):409-16. doi: 10.1016/j.ctim.2012.07.002. Epub 2012 Aug 23. PMID 23131371
- [Background] Licht CM, de Geus EJ, van Dyck R, Penninx BW. Association between anxiety disorders and heart rate variability in The Netherlands Study of Depression and Anxiety (NESDA). Psychosom Med. 2009 Jun;71(5):508-18. doi: 10.1097/PSY.0b013e3181a292a6. Epub 2009 May 4. PMID 19414616
- [Background] Luque-Casado A, Perakakis P, Ciria LF, Sanabria D. Transient autonomic responses during sustained attention in high and low fit young adults. Sci Rep. 2016 Jun 8;6:27556. doi: 10.1038/srep27556. PMID 27271980
- [Background] Mantella RC, Butters MA, Amico JA, Mazumdar S, Rollman BL, Begley AE, Reynolds CF, Lenze EJ. Salivary cortisol is associated with diagnosis and severity of late-life generalized anxiety disorder. Psychoneuroendocrinology. 2008 Jul;33(6):773-81. doi: 10.1016/j.psyneuen.2008.03.002. Epub 2008 Apr 14. PMID 18407426
- [Background] McConnell PA, Froeliger B, Garland EL, Ives JC, Sforzo GA. Auditory driving of the autonomic nervous system: Listening to theta-frequency binaural beats post-exercise increases parasympathetic activation and sympathetic withdrawal. Front Psychol. 2014 Nov 14;5:1248. doi: 10.3389/fpsyg.2014.01248. eCollection 2014. PMID 25452734
- [Background] Padmanabhan R, Hildreth AJ, Laws D. A prospective, randomised, controlled study examining binaural beat audio and pre-operative anxiety in patients undergoing general anaesthesia for day case surgery. Anaesthesia. 2005 Sep;60(9):874-7. doi: 10.1111/j.1365-2044.2005.04287.x. PMID 16115248
- [Background] Pittig A, Arch JJ, Lam CW, Craske MG. Heart rate and heart rate variability in panic, social anxiety, obsessive-compulsive, and generalized anxiety disorders at baseline and in response to relaxation and hyperventilation. Int J Psychophysiol. 2013 Jan;87(1):19-27. doi: 10.1016/j.ijpsycho.2012.10.012. Epub 2012 Oct 27. PMID 23107994
- [Background] Reedijk SA, Bolders A, Hommel B. The impact of binaural beats on creativity. Front Hum Neurosci. 2013 Nov 14;7:786. doi: 10.3389/fnhum.2013.00786. eCollection 2013. PMID 24294202
- [Background] Reedijk SA, Bolders A, Colzato LS, Hommel B. Eliminating the Attentional Blink through Binaural Beats: A Case for Tailored Cognitive Enhancement. Front Psychiatry. 2015 Jun 4;6:82. doi: 10.3389/fpsyt.2015.00082. eCollection 2015. PMID 26089802
- [Background] Roberts KE, Hart TA, Eastwood JD. Factor structure and validity of the State-Trait Inventory for Cognitive and Somatic Anxiety. Psychol Assess. 2016 Feb;28(2):134-146. doi: 10.1037/pas0000155. Epub 2015 May 25. PMID 26011481
- [Background] Tarrant J, Viczko J, Cope H. Virtual Reality for Anxiety Reduction Demonstrated by Quantitative EEG: A Pilot Study. Front Psychol. 2018 Jul 24;9:1280. doi: 10.3389/fpsyg.2018.01280. eCollection 2018. PMID 30087642
- [Background] Vedhara K, Miles J, Bennett P, Plummer S, Tallon D, Brooks E, Gale L, Munnoch K, Schreiber-Kounine C, Fowler C, Lightman S, Sammon A, Rayter Z, Farndon J. An investigation into the relationship between salivary cortisol, stress, anxiety and depression. Biol Psychol. 2003 Feb;62(2):89-96. doi: 10.1016/s0301-0511(02)00128-x. PMID 12581685
- [Background] Vreeburg SA, Zitman FG, van Pelt J, Derijk RH, Verhagen JC, van Dyck R, Hoogendijk WJ, Smit JH, Penninx BW. Salivary cortisol levels in persons with and without different anxiety disorders. Psychosom Med. 2010 May;72(4):340-7. doi: 10.1097/PSY.0b013e3181d2f0c8. Epub 2010 Feb 26. PMID 20190128
- [Background] Wahbeh H, Calabrese C, Zwickey H. Binaural beat technology in humans: a pilot study to assess psychologic and physiologic effects. J Altern Complement Med. 2007 Jan-Feb;13(1):25-32. doi: 10.1089/acm.2006.6196. PMID 17309374
- [Background] Watson D, Clark LA, Tellegen A. Development and validation of brief measures of positive and negative affect: the PANAS scales. J Pers Soc Psychol. 1988 Jun;54(6):1063-70. doi: 10.1037//0022-3514.54.6.1063. PMID 3397865
- [Derived] Ueberholz R, Glassman H, Mallik A, Russo FA. Effectiveness of music with auditory beat stimulation in reducing state anxiety in Canadian students with trait anxiety: protocol for a randomised controlled trial. BMJ Open. 2025 Jun 17;15(6):e094784. doi: 10.1136/bmjopen-2024-094784. PMID 40527557